CLINICAL TRIAL: NCT01299272
Title: LY2216684 Compared to Placebo as Adjunctive Therapy to SSRI in the Prevention of Symptom Re-emergence in Major Depressive Disorder
Brief Title: A Study in Prevention of Re-emergence of Depression Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11317; H9P-MC-LNBN (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2216684 + SSRI (Experimental): Acute Open-label (OL) Period: Participants received a starting dose of 12 milligrams (mg) LY2216684, administered orally, once daily for at least 2 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). Then, based on efficacy and tolerability, the dose could be increased to 18 mg (and decreased back to 12 mg) over the next 6 weeks.
  Stabilization OL Period: Participants meeting remission criteria continued on the same dose of LY2216684 for an additional 12 weeks. Participants who discontinued early during either OL Period were discontinued abruptly from LY2216684.
  Double-blind (DB) Randomized Withdrawal Period: At 20 weeks, participants meeting criteria for randomization continued their current dose of LY2216684 for another 24 weeks. Participants who completed this period or discontinued early were randomized to abrupt (placebo for 2 weeks) or tapered (12 mg LY2216684 for 4 days, 6 mg LY2216684 for 4 days, then placebo for 6 days) discontinuation of LY2216684.
  Interventions: Drug: LY2216684; Drug: SSRI
- Placebo + SSRI (Placebo Comparator): Acute Open-label (OL) Period: Participants received a starting dose of 12 milligrams (mg) LY2216684, administered orally, once daily for at least 2 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). Then, based on efficacy and tolerability, the dose could be increased to 18 mg (and decreased back to 12 mg) over the next 6 weeks.
  Stabilization OL Period: Participants meeting remission criteria continued on the same dose of LY2216684 for an additional 12 weeks. Participants who discontinued early during either OL Period were discontinued abruptly from LY2216684.
  Double-blind (DB) Randomized Withdrawal Period: At 20 weeks, participants meeting criteria for randomization were tapered from their LY2216684 dose to placebo following the regimen of 12 mg for 7 days, 6 mg for 7 days, and placebo for the remaining 22 weeks. Participants who completed this period or discontinued early continued to receive placebo for an additional 2 weeks
  Interventions: Drug: LY2216684; Drug: Placebo; Drug: SSRI

INTERVENTIONS:
Drug: LY2216684
  Other Names: Edivoxetine
Drug: Placebo
  Arms: Placebo + SSRI
Drug: SSRI — Participants should have been on their SSRI for at least 8 weeks prior and were to continue on their stable dose throughout the study.
  Other Names: Selective Serotonin Reuptake Inhibitor

SUMMARY:
The primary objective of this study was to assess the maintenance of efficacy of LY2216684 compared with placebo as adjunctive therapy to selective serotonin reuptake inhibitors (SSRIs) as measured by the time-to-symptom reemergence among participants with major depressive disorder (MDD) who met randomization criteria with adjunctive LY2216684 during the stabilization period.

This trial consists of two distinct periods: an open-label treatment period, which consists of two parts, 8 weeks acute open-label with movement to 12 weeks open-label stabilization if participants are in remission at end of 8 weeks (open-label for 20 weeks total) followed by a randomized, double-blind, placebo-controlled period for 24 weeks.

DETAILED DESCRIPTION:
In order to enter the Stabilization Open-label Period, participants must have met remission criteria, defined as a Montgomery-Asberg Depression Rating Scale (MADRS) total score ≤10 at Week 8. In order to enter the Double-blind Randomization Withdrawal Period, participants must have met randomization criteria, defined as a MADRS total score ≤10 at Weeks 18, 19, and 20.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with clinical diagnosis of Major Depressive Disorder (MDD)
* Using a reliable method of birth control
* Are taking a selective serotonin reuptake inhibitor (SSRI) approved for MDD treatment within the participant's country and the SSRI prescribed, including dose, should be consistent with labeling guidelines within the participating country
* Have a partial response to SSRI treatment
* Meet inclusion scores on pre-defined psychiatric scales to assess diagnosis of depression, disease severity, and response to SSRI treatment
* Reliable and able to keep all scheduled appointments
* Have had at least 1 previous episode of MDD prior to the current episode within the past 5 years

Exclusion Criteria:

* Have had or currently have any additional ongoing Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) Axis 1 condition other than major depression within 1 year of screening
* Have a current or any previous diagnosis of a bipolar disorder, schizophrenia, or other psychotic disorder
* Have a history of substance abuse and/or dependence within the past 1 year (drug categories defined by DSM-IV-TR), not including caffeine and nicotine.
* Have a DSM-IV-TR Axis II disorder that, in the judgment of the investigator, would interfere with compliance with protocol
* Have any diagnosed medical condition which could be exacerbated by noradrenergic agents, including unstable hypertension, unstable heart disease, tachycardia, tachyarrhythmia, narrow-angle glaucoma, or history of urinary hesitation or retention
* Have initiated or discontinued hormone therapy (including birth control or thyroid hormone) within the previous 3 months prior to enrollment
* Have a lifetime history of vagal nerve stimulation (VNS), transcranial magnetic stimulation (TMS), or psychosurgery
* Have received electroconvulsive therapy (ECT) in the past year
* Have a serious or unstable medical condition
* Have a history of seizure disorders
* Have initiated psychotherapy, change in intensity of psychotherapy or other nondrug therapies (such as acupuncture or hypnosis) within 6 weeks prior to enrollment or any time during the study
* Participants who, in the opinion of the investigator, are judged to be at serious risk for harm to self or others
* Are pregnant or breastfeeding
* Meet criteria for treatment-resistant depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1249 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (77):
- United States (27):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redlands, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherman Oaks, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Gables, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lafayette, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Terre Haute, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prairie Village, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clinton, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleton, Wisconsin
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Plata
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heusden-Zolder, Belgium
- Croatia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Split
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zagreb
- France (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arcachon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dole
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Douai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Élancourt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fains
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oranienburg
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haidari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tripoli
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camaiore-Viareggio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colleferro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ferrara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fracc. Bosques Del Prado Norte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Focşani
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
- Russia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Smolensk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stavropol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tomsk
- Slovakia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Banská Bystrica
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bratislava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Svidník
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zvolen
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salamanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Turkey (Türkiye) (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Adapazarı
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Diyarbakır

REFERENCES:
- [Derived] Oakes TM, Dellva MA, Waterman K, Greenbaum M, Poppe C, Goldberger C, Ahl J, Perahia DG. Edivoxetine compared to placebo as adjunctive therapy to selective serotonin reuptake inhibitors in the prevention of symptom re-emergence in major depressive disorder. Curr Med Res Opin. 2015 Jun;31(6):1179-89. doi: 10.1185/03007995.2015.1037732. Epub 2015 May 6. PMID 25894953

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants entered the Acute Open-label (OL) Period. At Week 8, if remission criteria were met, participants entered the Stabilization OL Period. At Week 20, if randomization criteria were met, participants entered the 24-week Double-blind Randomized Withdrawal Period. Those who discontinued early entered the Discontinuation Period.
Groups:
- LY2216684 + SSRI (Acute Open-label Period): Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
- LY2216684 + SSRI (Stabilization Open-label Period): Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD for an additional 12 weeks.
- LY2216684 + SSRI (Double-blind Randomized Withdrawal Period): Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD, for 12 weeks. At 20 weeks, participants meeting criteria for randomization continued at their current dose of LY2216684 and SSRI, orally, QD, for an additional 24 weeks.
- Placebo + SSRI (Double-blind Randomized Withdrawal Period): Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD, for 12 weeks. At 20 weeks, participants meeting criteria for randomization were switched from LY2216684 to Placebo and continued at their current SSRI dose, orally, QD, for an additional 24 weeks.
Period: Acute Open-label (OL) Period
Arm/Group | LY2216684 + SSRI (Acute Open-label Period) | LY2216684 + SSRI (Stabilization Open-label Period) | LY2216684 + SSRI (Double-blind Randomized Withdrawal Period) | Placebo + SSRI (Double-blind Randomized Withdrawal Period)
Started | 1249 | 0 | 0 | 0
Entered Discontinuation (DC) Period | 271 (Participants who discontinued the Acute OL Period had the option to enter the DC Period.) | 0 | 0 | 0
Completed | 835 (Participants who completed the Acute OL Period entered the Stabilization OL Period.) | 0 | 0 | 0
Not Completed | 414 | 0 | 0 | 0
Not completed — Remission Criteria Not Met | 140 | 0 | 0 | 0
Not completed — Adverse Event | 140 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 56 | 0 | 0 | 0
Not completed — Protocol Violation | 36 | 0 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0 | 0
Not completed — Sponsor Decision | 13 | 0 | 0 | 0
Not completed — Lack of Efficacy | 10 | 0 | 0 | 0
Not completed — Physician Decision | 5 | 0 | 0 | 0
Period: Stabilization Open-label (OL) Period
Arm/Group | LY2216684 + SSRI (Acute Open-label Period) | LY2216684 + SSRI (Stabilization Open-label Period) | LY2216684 + SSRI (Double-blind Randomized Withdrawal Period) | Placebo + SSRI (Double-blind Randomized Withdrawal Period)
Started | 0 | 835 | 0 | 0
Entered Discontinuation (DC) Period | 0 | 164 (Participants who discontinued the Stabilization OL Period had the option to enter the DC Period.) | 0 | 0
Completed | 0 | 586 (Participants who completed the Stabilization OL Period were randomized to the DB Period.) | 0 | 0
Not Completed | 0 | 249 | 0 | 0
Not completed — Randomization Criteria Not Met | 0 | 80 | 0 | 0
Not completed — Protocol Violation | 0 | 44 | 0 | 0
Not completed — Adverse Event | 0 | 42 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 42 | 0 | 0
Not completed — Sponsor Decision | 0 | 12 | 0 | 0
Not completed — Lack of Efficacy | 0 | 11 | 0 | 0
Not completed — Lost to Follow-up | 0 | 9 | 0 | 0
Not completed — Reemergence of Study Condition Symptoms | 0 | 6 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 0 | 0
Period: Double-blind (DB) Randomized Period
Arm/Group | LY2216684 + SSRI (Acute Open-label Period) | LY2216684 + SSRI (Stabilization Open-label Period) | LY2216684 + SSRI (Double-blind Randomized Withdrawal Period) | Placebo + SSRI (Double-blind Randomized Withdrawal Period)
Started | 0 | 0 | 294 | 292
Entered Taper Discontinuation Period | 0 | 0 | 129 (Participants who completed or discontinued the DB Period were randomized to the taper DC Period.) | 0
Entered Abrupt Discontinuation Period | 0 | 0 | 132 (Participants who completed or discontinued the DB Period were randomized to the abrupt DC Period.) | 268 (Participants who completed or discontinued the DB Period entered the DC Period.)
Completed | 0 | 0 | 224 | 234
Not Completed | 0 | 0 | 70 | 58
Not completed — Withdrawal by Subject | 0 | 0 | 22 | 15
Not completed — Lack of Efficacy | 0 | 0 | 20 | 10
Not completed — Adverse Event | 0 | 0 | 8 | 9
Not completed — Protocol Violation | 0 | 0 | 8 | 7
Not completed — Lost to Follow-up | 0 | 0 | 5 | 5
Not completed — Reemergence of Study Condition Symptoms | 0 | 0 | 4 | 10
Not completed — Physician Decision | 0 | 0 | 2 | 1
Not completed — Sponsor Decision | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- All Enrolled Participants: All enrolled participants started on a flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD, for an additional 12 weeks. At 20 weeks, participants meeting criteria for randomization either 1) continued at their current dose of LY2216684 and SSRI, orally, QD, for an additional 24 weeks or 2) were switched from LY2216684 to Placebo and continued at their current SSRI dose, orally, QD, for an additional 24 weeks.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1249
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 917
  Male | 332
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 50
  Asian | 21
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 99
  White | 1066
  More than one race | 13
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 254
  Not Hispanic or Latino | 622
  Unknown or Not Reported | 373
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 535
  Slovakia | 65
  Greece | 43
  Spain | 43
  Turkey | 30
  Russia | 96
  Italy | 44
  France | 61
  Mexico | 63
  Puerto Rico | 77
  Argentina | 62
  Belgium | 11
  Croatia | 9
  Romania | 19
  Germany | 73
  South Korea | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Meet Criteria for Re-emergence of Depressive Symptoms Estimated by Kaplan-Meier Product Limit Method (Double-blind Randomized Withdrawal Period)
Description: Participants meeting any of the following criteria were determined as having major depressive disorder symptom re-emergence: 1) a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater ≥14 or a Clinical Global Impressions of Severity (CGI-S) increase of 2 or more points from Week 18 at 2 consecutive visits or 2) discontinuation due to lack of efficacy/worsening of depression/suicidality. Time from randomization to the first visit at which the participant met the reemergence criteria was calculated. The percentage of participants who meet criteria was estimated using the Kaplan-Meier product limit method. The MADRS is a rating scale for severity of depressive mood symptoms and has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity) to 60 (high severity). CGI-S measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (extremely ill).
Time Frame: Randomization up to 44 weeks
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- LY2216684 + SSRI: Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD, for 12 weeks. At 20 weeks, participants meeting criteria for randomization continued at their current dose of LY2216684 and SSRI, orally, QD, for an additional 24 weeks.
- Placebo + SSRI: Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD, for 12 weeks. At 20 weeks, participants meeting criteria for randomization were switched from LY2216684 to Placebo and continued at their current SSRI dose, orally, QD, for an additional 24 weeks.
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 294 | 292
percentage of participants | 10.43 | 8.24
Statistical Analysis 1: Comparison: LY2216684 + SSRI vs Placebo + SSRI; Test type: Superiority or Other; p = 0.485, Log Rank

2. Secondary Outcome: Percentage of Participants With Re-emergence of Depressive Symptoms (Double-blind Randomized Withdrawal Period)
Description: Participants meeting any of the following criteria were determined as having major depressive disorder symptom re-emergence: 1) a Montgomery-Asberg Depression Rating Scale (MADRS) total score greater ≥14 or a Clinical Global Impressions of Severity (CGI-S) increase of 2 or more points from Week 18 at 2 consecutive visits or 2) discontinuation due to lack of efficacy/worsening of depression/suicidality. The percentage of participants with re-emergence of depressive symptoms was calculated by dividing the number of participants who meet any of the criteria by the total number of participants analyzed, multiplied by 100. The MADRS is a rating scale for severity of depressive mood symptoms and has a 10-item checklist with items rated on a scale of 0-6, for a total score range of 0 (low severity) to 60 (high severity). CGI-S measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (extremely ill).
Time Frame: Week 44
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 294 | 292
percentage of participants | 9.9 | 8.2

3. Secondary Outcome: Change From Randomization in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score and Individual Item Scores at Week 44 (Double-blind Randomized Withdrawal Period)
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which includes terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline MADRS total score (individual item score) and baseline MADRS total score (individual item score)-by-visit interaction.
Time Frame: Randomization, Week 44
Population: All randomized participants who have non-missing values at the time of randomization and at least one post-randomization value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 290 | 292
units on a scale
  MADRS Total Score | 0.40 (0.33) | 0.34 (0.33)
  Item 1: Apparent Sadness | 0.09 (0.05) | 0.08 (0.05)
  Item 2: Reported Sadness | 0.09 (0.06) | 0.05 (0.06)
  Item 3: Inner Tension | 0.06 (0.07) | 0.14 (0.06)
  Item 4: Reduced Sleep | -0.02 (0.07) | -0.06 (0.07)
  Item 5: Reduced Appetite | 0.00 (0.04) | -0.00 (0.04)
  Item 6: Concentration Difficulties | 0.07 (0.06) | 0.08 (0.06)
  Item 7: Lassitude | 0.02 (0.06) | 0.07 (0.06)
  Item 8: Inability to Feel | -0.00 (0.05) | -0.05 (0.05)
  Item 9: Pessimistic Thoughts | -0.01 (0.05) | -0.02 (0.04)
  Item 10: Suicidal Thoughts | 0.02 (0.02) | 0.01 (0.02)

4. Secondary Outcome: Change From Randomization in the Hospital Anxiety and Depression Scale (HADS) Depression and Anxiety Subscale Scores at Week 44 (Double-blind Randomized Withdrawal Period)
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a 'significant' case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal'. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline subscale score and baseline subscale score-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 286 | 285
units on a scale
  HADS Anxiety Subscale Score | -0.00 (0.22) | 0.15 (0.22)
  HADS Depression Subscale Score | -0.18 (0.23) | 0.15 (0.23)

5. Secondary Outcome: Change From Randomization in the Clinical Global Impression of Severity (CGI-S) Scores at Week 44 (Double-blind Randomized Withdrawal Period)
Description: The Clinical Global Impression of Severity (CGI-S) instrument is used to record the severity of mental illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline CGI-S score and baseline CGI-S score-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 290 | 292
units on a scale | 0.01 (0.05) | -0.00 (0.05)

6. Secondary Outcome: Change From Randomization in the Fatigue Associated With Depression (FAsD) Average Score, Experience Subscale Score, and Impact Subscale Score at Week 44 (Double-blind Randomized Withdrawal Period)
Description: The FAsD is a 13-item participant-rated scale. Items 1-6 ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Items 7-13 ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The experience subscale score is derived by taking the mean of Items 1-6. The impact subscale score is derived by taking the mean of applicable Items 7-13. The average score is the mean of applicable Items 1-13. Item 12 applies only to participants with a spouse or significant other and Item 13 applies to participants who had a job or who went to school. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 286 | 286
units on a scale
  FAsD Experience Subscale Score | -0.05 (0.05) | 0.05 (0.05)
  FAsD Impact Subscale Score | -0.06 (0.05) | -0.01 (0.05)
  FAsD Average Score | -0.05 (0.05) | 0.02 (0.05)

7. Secondary Outcome: Change From Randomization in the Sheehan Disability Scale (SDS) Items at Week 44 (Double-blind Randomized Withdrawal Period)
Description: The Sheehan Disability Scale (SDS) is completed by the participant and used to assess the effect of the participant's symptoms on their work (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline score and baseline score-by-visit interaction
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 289 | 289
units on a scale
  Work Impairment Score: number analyzed (Participants) | 198 | 212
  Work Impairment Score | -0.24 (0.17) | 0.02 (0.17)
  Social Life Impairment Score: number analyzed (Participants) | 286 | 286
  Social Life Impairment Score | -0.17 (0.14) | -0.15 (0.14)
  Family Life Impairment Score: number analyzed (Participants) | 286 | 286
  Family Life Impairment Score | -0.26 (0.14) | -0.08 (0.14)

8. Secondary Outcome: Change From Randomization in the EuroQol Questionnaire-5 Dimension (EQ-5D) Index Scores, Visual Analog Scale up to Week 44 (Double-blind Randomized Withdrawal Period)
Description: The EQ-5D, a health-related, quality-of-life instrument, contains 2 parts: a health status profile and a visual analog scale (VAS). The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3-level scale (no problem, some problems, and major problems). These dimensions are converted into weighted health-state index scores according to United States (US) and United Kingdom (UK) population-based algorithms. The US and UK based index scores range from -0.11 to 1.0 (where a score of 1.0 indicates perfect health) and from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension), respectively. The VAS consists of participants rating their current health state from 0 (worst imaginable health state) to 100 (best imaginable health). Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) model with main effects of treatment, country, and baseline score.
Time Frame: Randomization, up to Week 44
Population: All randomized participants who have non-missing values at the time of randomization and at least one post-randomization value. Last observation carried forward (LOCF) methodology was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 278 | 285
units on a scale
  EQ-5D US: number analyzed (Participants) | 278 | 284
  EQ-5D US | 0.01 (0.01) | 0.01 (0.01)
  EQ-5D UK: number analyzed (Participants) | 278 | 284
  EQ-5D UK | 0.01 (0.02) | 0.01 (0.02)
  VAS | 1.87 (1.39) | 0.61 (1.39)

9. Secondary Outcome: Number of Participants With Treatment-emergent Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) (Double-blind Randomized Withdrawal Period)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation is defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which includes a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation and behavior are defined as treatment-emergent (TE) if not present during the period up through randomization. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Randomization through Week 44
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 291 | 292
participants
  TE Suicidal Ideation | 5 | 4
  TE Suicidal Behavior: number analyzed (Participants) | 277 | 278
  TE Suicidal Behavior | 1 | 0

10. Secondary Outcome: Change From Randomization in the Arizona Sexual Experiences (ASEX) Questionnaire at Week 44 (Double-blind Randomized Withdrawal Period)
Description: Arizona Sexual Experiences (ASEX) Questionnaire is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Each item is rated from 1 (extremely) to 6 (no/never). Possible total scores ranged from 5 to 30, with the higher scores indicating more sexual dysfunction. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline ASEX total score and baseline ASEX total score-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 280 | 277
units on a scale | -0.39 (0.33) | -0.08 (0.33)

11. Secondary Outcome: Change From Randomization in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) Total Score at Week 44 (Double-blind Randomized Withdrawal Period)
Description: Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item is scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total score is reported and ranges from 7 to 42, with higher scores indicating greater impairment. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline CPFQ total score and baseline CPFQ total score-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 286 | 286
units on a scale | -0.27 (0.31) | -0.05 (0.31)

12. Secondary Outcome: Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score and Individual Item Scores up to Week 8 (Acute Open-label Period)
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline, up to Week 8
Population: All participants who have non-missing values at baseline and at least one post-baseline value. Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LY2216684 + SSRI: Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1214
units on a scale
  MADRS Total Score | -13.21 (8.30)
  Item 1: Apparent Sadness | -1.82 (1.37)
  Item 2: Reported Sadness | -1.86 (1.39)
  Item 3: Inner Tension | -1.24 (1.37)
  Item 4: Reduced Sleep | -1.29 (1.57)
  Item 5: Reduced Appetite | -0.65 (1.47)
  Item 6: Concentration Difficulties | -1.49 (1.43)
  Item 7: Lassitude | -1.74 (1.44)
  Item 8: Inability to Feel | -1.65 (1.42)
  Item 9: Pessimistic Thoughts | -1.23 (1.28)
  Item 10: Suicidal Thoughts | -0.24 (0.70)

13. Secondary Outcome: Change From Week 8 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score and Individual Item Scores up to Week 20 (Stabilization Open-label Period)
Description: as for outcome 12
Time Frame: Week 8, up to Week 20
Population: All participants who have non-missing values at Week 8 and at least one post-Week 8 value. Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LY2216684 + SSRI: Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI). At 8 weeks, participants meeting remission criteria continued on the same, stable dose of LY2216684 and SSRI, orally, QD for 12 weeks.
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 812
units on a scale
  MADRS Total Score | -0.38 (6.09)
  Item 1: Apparent Sadness | -0.01 (1.01)
  Item 2: Reported Sadness | -0.08 (1.15)
  Item 3: Inner Tension | -0.05 (1.18)
  Item 4: Reduced Sleep | -0.12 (1.28)
  Item 5: Reduced Appetite | 0.00 (0.89)
  Item 6: Concentration Difficulties | -0.06 (1.19)
  Item 7: Lassitude | 0.02 (1.19)
  Item 8: Inability to Feel | -0.09 (1.08)
  Item 9: Pessimistic Thoughts | -0.04 (0.87)
  Item 10: Suicidal Thoughts | 0.03 (0.47)

14. Secondary Outcome: Change From Baseline in the Hospital Anxiety and Depression Scale (HADS) Depression and Anxiety Subscale Scores up to Week 8 (Acute Open-label Period)
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale were considered to be a 'significant' case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal'.
Time Frame: Baseline, up to Week 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1199
units on a scale
  HADS Anxiety Subscale Score: number analyzed (Participants) | 1198
  HADS Anxiety Subscale Score | -3.02 (3.92)
  HADS Depression Subscale Score | -3.98 (4.41)

15. Secondary Outcome: Change From Week 8 in the Hospital Anxiety and Depression Scale (HADS) Depression and Anxiety Subscale Scores up to Week 20 (Stabilization Open-label Period)
Description: The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item is rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression. Scores of 11 or more on either subscale are considered to be a 'significant' case of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal'.
Time Frame: Week 8, up to Week 20
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 781
units on a scale
  HADS Anxiety Subscale Score | -0.77 (3.73)
  HADS Depression Subscale Score | -0.74 (3.57)

16. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity (CGI-S) Scores up to Week 8 (Acute Open-label Period)
Description: The Clinical Global Impression of Severity (CGI-S) instrument is used to record the severity of mental illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants).
Time Frame: Baseline, up to Week 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1214
units on a scale | -1.51 (1.17)

17. Secondary Outcome: Change From Week 8 in the Clinical Global Impression of Severity (CGI-S) Scores up to Week 20 (Stabilization Open-label Period)
Description: as for outcome 16
Time Frame: Week 8, up to Week 20
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 812
units on a scale | -0.25 (0.95)

18. Secondary Outcome: Change From Baseline in the Fatigue Associated With Depression (FAsD) Average Score, Experience Subscale Score, and Impact Subscale Score up to Week 8 (Acute Open-label Period)
Description: The Fatigue Associated With Depression (FAsD) is a 13-item participant-rated scale. Items 1-6 ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Items 7-13 ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The experience subscale score is derived by taking the mean of Items 1-6. The impact subscale score is derived by taking the mean of applicable Items 7-13. The average score is the mean of applicable Items 1-13. Item 12 applies only to participants with a spouse or significant other and Item 13 applies to participants who had a job or who went to school.
Time Frame: Baseline, up to Week 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1166
units on a scale
  FAsD Experience Subscale Score | -0.82 (0.99)
  FAsD Impact Subscale Score: number analyzed (Participants) | 1164
  FAsD Impact Subscale Score | -0.88 (1.03)
  FAsD Average Score: number analyzed (Participants) | 1164
  FAsD Average Score | -0.85 (0.93)

19. Secondary Outcome: Change From Week 8 in the Fatigue Associated With Depression (FAsD) Average Score, Experience Subscale Score, and Impact Subscale Score up to Week 20 (Stabilization Open-label Period)
Description: as for outcome 18
Time Frame: Week 8, up to Week 20
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 781
units on a scale
  FAsD Experience Subscale Score | -0.22 (0.93)
  FAsD Impact Subscale Score | -0.15 (0.87)
  FAsD Average Score | -0.19 (0.84)

20. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Items up to Week 8 (Acute Open-label Period)
Description: The Sheehan Disability Scale (SDS) is completed by the participant and used to assess the effect of the participant's symptoms on their work (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption.
Time Frame: Baseline, up to Week 8
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1197
units on a scale
  Work Impairment Score: number analyzed (Participants) | 757
  Work Impairment Score | -2.17 (2.65)
  Social Life Impairment Score | -2.38 (2.85)
  Family Life Impairment Score | -2.16 (2.81)

21. Secondary Outcome: Change From Week 8 in the Sheehan Disability Scale (SDS) Items up to Week 20 (Stabilization Open-label Period)
Description: as for outcome 20
Time Frame: Week 8, up to Week 20
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 781
units on a scale
  Work Impairment Score: number analyzed (Participants) | 567
  Work Impairment Score | -0.58 (2.61)
  Social Life Impairment Score | -0.47 (2.54)
  Family Life Impairment Score | -0.50 (2.50)

22. Secondary Outcome: Change From Baseline in the EuroQol Questionnaire-5 Dimension (EQ-5D) Index Scores, Visual Analog Scale up to Week 20 (Open-label Period)
Description: The EQ-5D, a health-related, quality-of-life instrument, contains 2 parts: a health status profile and a visual analog scale (VAS). The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a 3-level scale (no problem, some problems, and major problems). These dimensions are converted into weighted health-state index scores according to United States (US) and United Kingdom (UK) population-based algorithms. The US and UK based index scores range from -0.11 to 1.0 (where a score of 1.0 indicates perfect health) and from -0.59 (severe problems in all 5 dimensions) to 1.0 (no problem in any dimension), respectively. The VAS consists of participants rating their current health state from 0 (worst imaginable health state) to 100 (best imaginable health).
Time Frame: Baseline, up to Week 20
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 779
units on a scale
  EQ-5D US: number analyzed (Participants) | 773
  EQ-5D US | 0.15 (0.19)
  EQ-5D UK: number analyzed (Participants) | 773
  EQ-5D UK | 0.21 (0.29)
  VAS | 18.07 (22.15)

23. Secondary Outcome: Number of Participants With Treatment-emergent Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) (Open-label Period)
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation is defined as a "yes" answer to any 1 of 5 suicidal ideation questions, which included a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation and behavior are defined as treatment-emergent (TE) if not present at baseline. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Baseline through Week 20
Population: All participants who have non-missing values at baseline and at least one post-baseline value.
Measure: Number; unit: participants
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1216
participants
  TE Suicidal Ideation | 66
  TE Suicidal Behavior: number analyzed (Participants) | 1124
  TE Suicidal Behavior | 5

24. Secondary Outcome: Change From Baseline in the Arizona Sexual Experiences (ASEX) Questionnaire up to Week 20 (Open-label Period)
Description: Arizona Sexual Experiences (ASEX) Questionnaire is a 5-item rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. Each item is rated from 1 (extremely) to 6 (no/never). Possible total scores ranged from 5 to 30, with the higher scores indicating more sexual dysfunction.
Time Frame: Baseline, up to Week 20
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1115
units on a scale | -1.78 (4.98)

25. Secondary Outcome: Change From Baseline in the Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) Total Score at Week 20 (Open-label Period)
Description: Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ) is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item is scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total score is reported and ranges from 7 to 42, with higher scores indicating greater impairment.
Time Frame: Baseline, up to Week 20
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1167
units on a scale | -6.68 (7.03)

26. Secondary Outcome: Change From Randomization in Blood Pressure at Week 44 (Double-blind Randomized Withdrawal Period)
Description: Blood pressure measurements were taken 3 times at each visit in a sitting position. The average of the 3 values was used for analysis. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline and baseline-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 291 | 292
millimeters of mercury (mmHg)
  Systolic blood pressure | -0.20 (0.75) | -4.19 (0.75)
  Diastolic blood pressure | 0.24 (0.55) | -4.18 (0.55)

27. Secondary Outcome: Change From Baseline in Blood Pressure up to Week 20 (Open-label Period)
Description: Blood pressure measurements were taken 3 times at each visit in a sitting position. The average of the 3 values was used for analysis.
Time Frame: Baseline, up to Week 20
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1214
millimeters of mercury (mmHg)
  Systolic blood pressure | 2.30 (11.95)
  Diastolic blood pressure | 2.81 (8.63)

28. Secondary Outcome: Change From Randomization in Pulse Rate at Week 44 (Double-blind Randomized Withdrawal Period)
Description: Pulse rate measurements were collected when the participant was in a sitting position. Least Squares (LS) means were calculated using a mixed model repeated measures (MMRM) analysis which included terms for the fixed categorical effects of treatment, country, visit, and treatment-by-visit interaction, as well as the continuous, fixed covariates of baseline and baseline-by-visit interaction.
Time Frame: Randomization, Week 44
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 291 | 292
beats per minute (bpm) | -2.54 (0.74) | -10.76 (0.74)

29. Secondary Outcome: Change From Baseline in Pulse Rate up to Week 20 (Open-label Period)
Description: Pulse measurements were collected when the participant was in a sitting position.
Time Frame: Baseline, up to Week 20
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 1214
beats per minute (bpm) | 10.80 (12.47)

ADVERSE EVENTS:
Groups:
- LY2216684 + SSRI (Acute Open-label Period): Flexible dose of 12 or 18 milligrams (mg) LY2216684, administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes all enrolled participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-baseline visit during the Acute Open-label Period.
- LY2216684 + SSRI (Stabilization Open-label Period): Same, stable dose of LY2216684 as in the Acute Open-label Period, orally, once daily (QD) for 12 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes all participants who completed the Acute Open-label Period and did not discontinue for the reason 'Lost to Follow-up' at the first post-baseline visit during the Stabilization Open-label Period.
- LY2216684 + SSRI (Double-blind Randomized Withdrawal Period): Same, stable dose of LY2216684 as in the Stabilization Open-label Period, orally, once daily (QD) for 24 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Double-blind Randomized Withdrawal Period.
- Placebo + SSRI (Double-blind Randomized Withdrawal Period): Placebo, orally, once daily (QD) for 24 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Double-blind Randomized Withdrawal Period.
- LY2216684 + SSRI (Randomized Tapered Discontinuation Period): 12 milligrams (mg) LY2216684 for 4 days, 6 mg LY2216684 for 4 days, then placebo for 6 days, orally, once daily (QD), adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes all randomized participants who tapered discontinuation of LY2216684 after completion of or early withdrawal from the Double-blind Randomized Withdrawal Period and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation Period visit.
- LY2216684 + SSRI (Randomized Abrupt Discontinuation Period): Placebo, orally, once daily (QD) for 2 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes all randomized participants who abruptly discontinued LY2216684 after completion of or early withdrawal from the Double-blind Randomized Withdrawal Period and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation Period visit.
- Placebo + SSRI (Abrupt Discontinuation Period): Placebo, orally, once daily (QD) for 2 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes all randomized participants who discontinued placebo after completion of or early withdrawal from the Double-blind Randomized Withdrawal Period and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation Period visit.
- LY2216684 + SSRI (Nonrandomized Abrupt Discontinuation Period): Placebo, orally, once daily (QD) for 2 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI).
  Includes all non-randomized participants who discontinued early from either Open-label Period and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation Period visit.
Arm/Group | LY2216684 + SSRI (Acute Open-label Period) | LY2216684 + SSRI (Stabilization Open-label Period) | LY2216684 + SSRI (Double-blind Randomized Withdrawal Period) | Placebo + SSRI (Double-blind Randomized Withdrawal Period) | LY2216684 + SSRI (Randomized Tapered Discontinuation Period) | LY2216684 + SSRI (Randomized Abrupt Discontinuation Period) | Placebo + SSRI (Abrupt Discontinuation Period) | LY2216684 + SSRI (Nonrandomized Abrupt Discontinuation Period)
Serious Adverse Events (participants affected / at risk) | 19/1244 | 15/831 | 2/294 | 6/292 | 2/128 | 0/132 | 2/267 | 8/434
Other Adverse Events (participants affected / at risk) | 505/1244 | 112/831 | 37/294 | 21/292 | 9/128 | 4/132 | 16/267 | 32/434
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2216684 + SSRI (Acute Open-label Period) (N=1244) | LY2216684 + SSRI (Stabilization Open-label Period) (N=831) | LY2216684 + SSRI (Double-blind Randomized Withdrawal Period) (N=294) | Placebo + SSRI (Double-blind Randomized Withdrawal Period) (N=292) | LY2216684 + SSRI (Randomized Tapered Discontinuation Period) (N=128) | LY2216684 + SSRI (Randomized Abrupt Discontinuation Period) (N=132) | Placebo + SSRI (Abrupt Discontinuation Period) (N=267) | LY2216684 + SSRI (Nonrandomized Abrupt Discontinuation Period) (N=434)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0/914 (0) | 1/641 (1) | 0/223 (0) | 0/226 (0) | 0/95 (0) | 0/105 (0) | 0/212 (0) | 0/307 (0)
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1/914 (1) | 0/641 (0) | 0/223 (0) | 0/226 (0) | 0/95 (0) | 0/105 (0) | 0/212 (0) | 1/307 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Self injurious behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal polyp (Reproductive system and breast disorders) | 0/914 (0) | 1/641 (1) | 1/223 (1) | 0/226 (0) | 0/95 (0) | 0/105 (0) | 0/212 (0) | 0/307 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0/914 (0) | 1/641 (1) | 0/223 (0) | 0/226 (0) | 0/95 (0) | 0/105 (0) | 0/212 (0) | 0/307 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2216684 + SSRI (Acute Open-label Period) (N=1244) | LY2216684 + SSRI (Stabilization Open-label Period) (N=831) | LY2216684 + SSRI (Double-blind Randomized Withdrawal Period) (N=294) | Placebo + SSRI (Double-blind Randomized Withdrawal Period) (N=292) | LY2216684 + SSRI (Randomized Tapered Discontinuation Period) (N=128) | LY2216684 + SSRI (Randomized Abrupt Discontinuation Period) (N=132) | Placebo + SSRI (Abrupt Discontinuation Period) (N=267) | LY2216684 + SSRI (Nonrandomized Abrupt Discontinuation Period) (N=434)
Constipation (Gastrointestinal disorders) | 132 (134) | 14 (14) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 80 (81) | 10 (10) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 147 (155) | 18 (21) | 7 (7) | 5 (5) | 3 (3) | 1 (1) | 5 (6) | 8 (10)
Dizziness (Nervous system disorders) | 83 (86) | 8 (8) | 3 (3) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 111 (128) | 53 (54) | 18 (24) | 13 (13) | 7 (10) | 4 (5) | 11 (16) | 24 (30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 215 (228) | 23 (24) | 8 (8) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days